CLINICAL TRIAL: NCT00292110
Title: Treatment of Heroin and Cocaine With Methadone Maintenance and Contingency Management
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 999904390; 04-DA-N390
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-08-09

CONDITIONS: Opiate-Related Disorders; Cocaine-Related Disorders
Keywords: HIV; Opiate Substitution; Pharmacokinetics; ECG; Polydrug Abuse
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Methadone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Arm Four (Active Comparator)
  Interventions: Drug: Methadone; Behavioral: Contingency Management/Noncontingent Incentives
- Arm One (Experimental)
  Interventions: Behavioral: Contingency Management; Drug: Methadone dose
- Arm Three (Active Comparator)
  Interventions: Drug: Methadone dose
- ArmTwo (Active Comparator)
  Interventions: Drug: Methadone; Behavioral: Contingency Management; Behavioral: Contingency Management/Noncontingent Incentives

INTERVENTIONS:
Drug: Methadone — 100 mg/day orally
  Arms: Arm Four; ArmTwo
Behavioral: Contingency Management — Incentives given for cocaine abstinence
  Arms: Arm One; ArmTwo
Drug: Methadone dose — flexible methadone dosing to 190 mg/day daily orally
  Arms: Arm One; Arm Three
Behavioral: Contingency Management/Noncontingent Incentives — Incentives given independent of drug use
  Arms: Arm Four; ArmTwo

SUMMARY:
Background:

- The treatment of addiction often hinges on preventing relapse into drug-using behaviors, which occurs at high rates even after prolonged abstinence. Some methadone patients continue to abuse cocaine and heroin during treatment, even with extensive psychosocial services. More research is needed to look at the results from earlier studies of continued drug use during methadone treatment, focusing on the results of fixed vs. flexible doses of methadone to reduce the likelihood of continued drug use and the role of monetary vouchers as an incentive to continue abstinence from illicit substances.

Objectives:

- To determine if the combination of flexible methadone dosing and voucher-based contingency management can improve rates of abstinence from heroin and cocaine.

Eligibility:

- Individuals between 18 and 65 years of age or older who are dependent on opioids (cocaine and/or heroin).

Design:

* The study will last 40 weeks. After the initial screening, participants will receive daily methadone and weekly drug counseling sessions that will continue throughout the study.
* After 6 weeks of methadone treatment, participants who continue to use heroin and cocaine will be randomized to one of four groups for 16 weeks of study. Each group will receive a flexible or fixed dose of methadone, and one of two contingency management conditions.
* Flexible-dose participants will receive individualized dose increases, based on drug use and withdrawal. Fixed-dose participants will be set at a specific dose of methadone that will not be changed.
* The two contingency management conditions will be monetary vouchers given for regular cocaine-negative urine samples, or vouchers independent of urine cocaine screen results.
* After the study phase, participants will have 10 weeks of standard individual counseling and stable doses of methadone. Urine samples will continue to be collected, but no vouchers will be given.
* At the end of the study, participants will have the choice of transferring to a community clinic or undergoing a 10-week taper from methadone.

DETAILED DESCRIPTION:
Scientific goals. The primary goal is to determine if simultaneous abstinence from heroin and cocaine can be elicited by combining two approaches: flexible methadone dosing and voucher-based CM. Secondary goals include: 1) comparing saliva and plasma levels of methadone, cortisol, and prolactin as predictors of treatment outcome; and 2) evaluating the impact of methadone maintenance on renal function, lipid profile, and cardiac function.

Methods. During an initial 6-week baseline phase, cocaine-abusing opioid-dependent outpatient participants (300 enrolled; 180 evaluable) will be stabilized on methadone 70 mg/day. At the end of baseline, participants who continue to use heroin and cocaine will be randomized to one of two dosing regimens and one of two CM conditions. In the flexible-dose regimen, participants will receive individualized dose increases (15 mg/day) to a maximum of 190 mg /day, based on heroin use and withdrawal. In the fixed-dose regimen, participants methadone dose will be increased to 100 mg/day and remain fixed there. Dose-group assignment will be double-blind: investigators will determine participants individualized dose increases, but only the pharmacists will know which participants actually receive them. The two CM conditions will be: vouchers contingent on cocaine-negative urine specimens, or noncontingent vouchers (i.e., vouchers independent of urine cocaine screen results). The main outcome measure will be the percentage of urines simultaneously negative for both cocaine and illicit opiates during treatment. For the concurrently run pharmacokinetic-pharmacodynamic portion, saliva and blood samples will be taken at regular intervals to determine levels of methadone, cortisol, and prolactin as predictors of treatment outcome. For the concurrently run medical-outcomes portion, urine (renal function), blood (lipid profile), and ECGs (cardiac function),will be obtained at set intervals.

Hypothesis. Flexible methadone dosing and voucher-based CM will be safe and result in greater simultaneous abstinence from heroin and cocaine, higher treatment retention, and higher health-related QOL when compared to fixed methadone dosing and the absence of CM.

Benefits. Participants will receive methadone, counseling, and some medical care at no charge. The methadone and voucher interventions are likely to reduce participants' use of heroin and cocaine. Counseling will include management of HIV risk behaviors. The study incorporates participant safety monitoring and will provide information relevant to improving the health and safety of community methadone-maintenance patients. The pharmacokinetic-pharmacodynamic part of the study does not benefit participants directly, but may lead to the development of more useful and less invasive drug-monitoring methods.

Risks. Participants may experience side effects from methadone, discomfort during methadone withdrawal, and discomfort (or, rarely syncope) from blood draws.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. age between 18 and 65;
  2. physical dependence on opioids
  3. evidence of cocaine use, by urine screen and self-report
  4. able to attend methadone clinic 7 days/week

EXCLUSION CRITERIA:

1. History of schizophrenia or any other DSM-IV psychotic disorder
2. History of bipolar disorder
3. Current Major Depressive Disorder;
4. Current physical dependence on alcohol or sedative-hypnotics, e.g. benzodiazepines
5. Cognitive impairment severe enough to preclude informed consent or valid responses on questionnaires (Shipley Institute of Living scale-estimated full-scale IQ less than 80)
6. Medical illness that in the view of the investigators would compromise participation in research
7. Urologic conditions that would inhibit urine collection
8. Previous bowel obstruction.
9. Previous history of the following: major abdominal surgery, major gynecologic / pelvic surgery, inflammatory bowel disease (Crohn s or ulcerative colitis), Meckel s diverticulum, congenital atresia or stenosis, diverticulitis, radiation enteropathy or stricture, bowel neoplasm, endometriosis, inguinal-femoral-umbilical-ventral hernia, volvulus, or neurogenic megacolon, frequent bezoars.
10. Recent use of medications known to cause severe constipation.
11. History of previous severe respiratory depression or coma due to methadone use.
12. Pregnancy.
13. Personal history of a serious arrhythmia such as ventricular tachycardia, ventricular fibrillation, or Torsade de pointes; personal history of congenital heart disease or arrhythmia.
14. Personal history of congenital long QT syndrome (LQT).
15. Family history of a congenital long QT syndrome.
16. Family history of Torsade de pointes.
17. Family history of sudden cardiac death below the age of forty years.
18. Evidence of clinically significant structural heart disease.
19. Personal history of severe electrolyte disorders.
20. Recent use of anti-arrhythmic agents.
21. Poor venous access.
22. Lab values outside the parameters set in Table II. These exclusion values are based upon the Medical Screening guideline used previously at the NIDA-IRP.
23. CD4 less than 200 or evidence of severely compromised immune system / AIDS
24. Women who are able to get pregnant must agree to use a medically effective form of contraception while in the study.

Acceptable forms of contraception for this study include:

1. Hormonal contraception (birth control pills, injected hormones, vaginal ring)
2. Intrauterine device
3. Barrier methods with spermicide (diaphragm with spermicide, condom with spermicide)
4. Surgical sterilization (hysterectomy, tubal ligation, or vasectomy in a partner)

Women who do not agree to use these medically effective forms of contraception while in the study will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2004-02-01; Primary Completion 2013-08-09 (Actual); Study Completion 2013-08-09 (Actual)

PRIMARY OUTCOMES:
Abstinence from cocaine and heroin | 16 weeks

SECONDARY OUTCOMES:
Time to relapse | 24 weeks
Psychological and psychosocial outcome | 50 weeks
HIV Risk Behaviors | 50 weeks
QT interval | 24 weeks
Urine microalbuminuria | 24 weeks
Blood lipid profile | 50 weeks
Quality of life | 50 weeks
Substance Dependence | 50 weeks
Methadone plasma and saliva concentration | 50 weeks
Cortisol and prolactin levels | 50 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kenzie Preston, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

REFERENCES:
- [Background] Ball JC, Lange WR, Myers CP, Friedman SR. Reducing the risk of AIDS through methadone maintenance treatment. J Health Soc Behav. 1988 Sep;29(3):214-26. No abstract available. PMID 3241064
- [Background] Barthwell A, Senay E, Marks R, White R. Patients successfully maintained with methadone escaped human immunodeficiency virus infection. Arch Gen Psychiatry. 1989 Oct;46(10):957-8. doi: 10.1001/archpsyc.1989.01810100099020. No abstract available. PMID 2802930
- [Background] Belding MA, McLellan AT, Zanis DA, Incmikoski R. Characterizing "nonresponsive" methadone patients. J Subst Abuse Treat. 1998 Nov-Dec;15(6):485-92. doi: 10.1016/s0740-5472(97)00292-4. PMID 9845861